CLINICAL TRIAL: NCT02908464
Title: Prevention of Early Postoperative Decline
Acronym: PEaPoD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Lumos Labs, Inc. (Industry)
Responsible Party: Principal Investigator, Brian O'Gara, MD, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016P000145
Record Dates: First submitted 2016-08-30; First posted 2016-09-21 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Delirium; Postoperative Cognitive Dysfunction
Keywords: Cardiac Surgery; Delirium; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Delirium; Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Lumosity (CT Group) (Experimental): Patients in the Lumosity arm will be prescribed a perioperative neurocognitive training program created in collaboration with Lumos Labs, Inc. The program will contain "brain games" that focus on enhancing cognitive abilities in working memory, attention, and processing speed. Participants will be expected to complete at least 2, but no more than 3, 15 minute sessions of training per day. The protocol will be prescribed for 10 days preoperatively, and then for four weeks postoperatively.
  Interventions: Device: Lumosity
- Usual Care (Control Group) (No Intervention): Patients in the usual care arm will undergo current standard of care for cardiac surgery and postoperative recovery. They will be asked to refrain from acquiring a Lumosity account.

INTERVENTIONS:
Device: Lumosity — A neurocognitive training program designed to enhance cognitive abilities
  Other Names: Brain Games
  Arms: Lumosity (CT Group)

SUMMARY:
The purpose of this trial is to determine whether using a brain training program in the time leading up to as well as after heart surgery will reduce confusion and cognitive loss that can occur after surgery.

DETAILED DESCRIPTION:
Randomized, controlled pilot study with a convenience sample of 45 adult cardiac surgical patients. The main intervention to be studied will be the use of a neurocognitive training program (Lumosity) for 10 days preoperatively, and then for four weeks postoperatively. The prescribed regimen of training will focus on the areas of cognitive function most commonly affected in the postoperative period, including working memory, attention, and processing speed. Patients in the control arm will undergo current standard cardiac surgical postoperative care and will be asked to refrain from obtaining a Lumosity account.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing cardiac surgery age 60-90
* Cardiac surgery scheduled at least 10 days from enrollment
* High school education level or equivalent

Exclusion Criteria:

* Preexisting psychiatric illness
* History of cerebrovascular event or seizure
* Non English speakers
* Baseline severe cognitive dysfunction including Alzheimer's, Parkinson's, or other severe forms of dementia
* Significant visual impairment
* Enrollment in another study involving cognition

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-11; Primary Completion 2019-01 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian O'Gara, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Gara B, Marcantonio ER, Pascual-Leone A, Shaefi S, Mueller A, Banner-Goodspeed V, Talmor D, Subramaniam B. Prevention of Early Postoperative Decline (PEaPoD): protocol for a randomized, controlled feasibility trial. Trials. 2018 Dec 11;19(1):676. doi: 10.1186/s13063-018-3063-z. PMID 30537982

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After participant enrollment, a baseline cognitive assessment was performed using the Montreal Cognitive Assessment (MoCA). If the patient achieved a score indicating the presence of severe baseline cognitive impairment (<10), they were subsequently withdrawn.
Period: Overall Study
Arm/Group | Lumosity (CT Group) | Usual Care (Control Group)
Started | 22 | 23
Completed | 20 | 20
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Found ineligible after randomization | 0 | 2

BASELINE CHARACTERISTICS:
Population: Among the 45 randomly assigned participants, 5 patients' participation was terminated and they were, therefore, excluded from subsequent analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumosity (CT Group) | Usual Care (Control Group) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (6) | 69 (7) | 70 (4.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 14 | 15 | 29
  Female | 6 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 19 | 19 | 38
  Race/Ethnicity: Black or African American | 0 | 0 | 0
  Race/Ethnicity: Asian | 1 | 0 | 1
  Race/Ethnicity: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race/Ethnicity: American Indian or Alaskan Native | 0 | 0 | 0
  Race/Ethnicity: Multi-Racial | 0 | 0 | 0
  Race/Ethnicity: Unknown | 0 | 0 | 0
  Race/Ethnicity: Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Language Status [Count of Participants; unit: Participants]
  Native born English speaker | 17 | 19 | 36
  Foreign born, English is second language | 3 | 1 | 4
Education Level [Count of Participants; unit: Participants]
  High school graduate or equivalent | 1 | 5 | 6
  Some college, associate's degree | 4 | 2 | 6
  Bachelor's degree | 8 | 5 | 13
  Master's degree | 5 | 4 | 9
  Doctoral degree | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Providing a Neurocognitive Training Program to Elderly Cardiac Surgical Patients - Enrollment
Description: Feasibility will be partly determined by evaluating enrollment. Enrolling >50% of eligible patients is the target.
Time Frame: Enrollment was assessed after enrollment was completed.
Population: This population is of patients who after screening met the eligibility criteria and were approached for this study. The total count of participants depict the total number enrolled.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study Enrollment: This group includes the enrollment of patients in the Lumosity arm (CT Group), as well as the patients in the usual care arm (Control Group).
Arm/Group | Overall Study Enrollment
Number analyzed (Participants) | 69
Participants | 45

2. Primary Outcome: Feasibility of Providing a Neurocognitive Training Program to Elderly Cardiac Surgical Patients - Adherence
Description: Feasibility will be partly determined by evaluating adherence patterns. Sufficient adherence to protocol will be deemed sufficient to deem the study feasible.
Time Frame: To be evaluated at the conclusion of the study. Adherence was assessed in 3 separate periods: pre hospital, in hospital, and post discharge (typically at the 4 week follow up clinic visit).
Measure: Median (Inter-Quartile Range); unit: percentage of minutes trained/prescribed
Arm/Group | Lumosity (CT Group) | Usual Care (Control Group)
Number analyzed (Participants) | 20 | 20
percentage of minutes trained/prescribed
  Pre-Hospital Training Adherence | 39 [20 to 68] | 0 [0 to 0]
  In-Hospital Training Adherence | 6 [0 to 37] | 0 [0 to 0]
  Post-Discharge Training Adherence | 19 [0 to 56] | 0 [0 to 0]

3. Secondary Outcome: Number of Participants With Postoperative Delirium Measured by the Confusion Assessment Method (CAM)
Description: Condition characterized by inattention and fluctuating consciousness. Measured by the Confusion Assessment Method (CAM).
  Inouye, S., van Dyck, C., Alessi, C., Balkin, S., Siegal, A. & Horwitz, R. (1990). Clarifying confusion: The confusion assessment method. Annals of Internal Medicine, 113(12), 941-948.
Time Frame: Defined as present or absent on any day from postoperative day 1 to postoperative day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Lumosity (CT Group) | Usual Care (Control Group)
Number analyzed (Participants) | 20 | 20
Participants
  Delrium present | 5 | 3
  Delirium not present | 15 | 17

4. Secondary Outcome: Number of Participants With Postoperative Cognitive Decline
Description: Condition characterized by decrease in cognitive performance by one standard deviation after surgery, as compared to baseline. Measured by the Montreal Cognitive Assessment (MoCA).
Time Frame: Day of hospital discharge, an average of 1 week.
Population: The discrepancy of participants analyzed comes from missed assessments due to unavailability of study staff.
Measure: Count of Participants; unit: Participants
Arm/Group | Lumosity (CT Group) | Usual Care (Control Group)
Number analyzed (Participants) | 17 | 19
Participants
  Cognitive decline present | 9 | 7
  Cognitive decline not present | 8 | 12

5. Secondary Outcome: Postoperative Cognitive Dysfunction Measured Using the Montreal Cognitive Assessment (MoCA)
Description: Condition characterized by loss of cognitive function after surgery.
  Measured using the telephonic Montreal Cognitive Assessment (t-MoCA). The minimum score is 0, the maximum score is 22. The higher the score, the better the outcome.
Time Frame: Measured at 1, 3 and 6 months postoperatively.
Population: The number analyzed decreases and increases at different time points due to the inconsistency of utilizing telephone calls to obtain cognitive scores, and the difficulty of reliably reaching patients.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Lumosity (CT Group) | Usual Care (Control Group)
Number analyzed (Participants) | 17 | 19
score on a scale
  Postoperative t-MoCA score (0-22, 22 best) Month 1 | 20.0 [18.0 to 21.0] | 19.0 [18.0 to 21.0]
  Postoperative t-MoCA score (0-22, 22 best) Month 3: number analyzed (Participants) | 11 | 13
  Postoperative t-MoCA score (0-22, 22 best) Month 3 | 20.0 [19.0 to 21.0] | 21.0 [20.0 to 21.0]
  Postoperative t-MoCA score (0-22, 22 best) Month 6: number analyzed (Participants) | 13 | 14
  Postoperative t-MoCA score (0-22, 22 best) Month 6 | 20.0 [19.0 to 22.0] | 20.5 [18.0 to 21.0]

6. Other Pre Specified Outcome: Postoperative Survey
Description: Satisfaction with CT was assessed postoperatively at the follow up visit. Survey questions were both structured and open-ended. Quantitative scales were used to assess the level of agreement with prompted statements, using slide bars with visible anchors of "strongly disagree" (0), "neutral" (50), and "strongly agree" (100). The final question was only asked of the control patients to gauge their theoretical interest in using cognitive training for a future surgery.
Time Frame: Postoperative visit (usually within 1 month after discharge)
Population: Complete study population
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Lumosity (CT Group) | Usual Care (Control Group)
Number analyzed (Participants) | 20 | 20
Scores on a scale
  The program was easy to use: number analyzed (Participants) | 20 | 0
  The program was easy to use | 87 [75 to 97] |
  I enjoyed playing the games: number analyzed (Participants) | 20 | 0
  I enjoyed playing the games | 85 [79 to 91] |
  I think my memory improved | 75 [54 to 82] | 51 [49 to 54]
  I think my thinking ability improved | 78 [64 to 83] | 50 [41 to 68]
  I would be interested in CT for another surgery: number analyzed (Participants) | 0 | 20
  I would be interested in CT for another surgery |  | 70 [50 to 86]

7. Other Pre Specified Outcome: Patient Satisfaction
Description: Overall satisfaction with participating in the study. Measured on a scale of 0-100 with higher values representing higher satisfaction.
Time Frame: Postoperative visit (usually within 1 month after discharge)
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Lumosity (CT Group) | Usual Care (Control Group)
Number analyzed (Participants) | 20 | 20
scores on a scale | 90 [78 to 94] | 74 [67 to 87]

8. Other Pre Specified Outcome: Postoperative Survey (Cont)
Description: A final question asked on the postoperative satisfaction survey: Preparation and recovery from cardiac surgery should include some form of brain training program. Results are count of participants answering yes.
Time Frame: Postoperative visit (usually within 1 month after discharge)
Population: Question not asked of the CT group participants
Measure: Count of Participants; unit: Participants
Arm/Group | Lumosity (CT Group) | Usual Care (Control Group)
Number analyzed (Participants) | 0 | 20
Participants |  | 17

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed through the 6 month follow up.
Arm/Group | Lumosity (CT Group) | Usual Care (Control Group)
All-Cause Mortality (participants affected / at risk) | 2/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT02908464/Prot_SAP_000.pdf